CLINICAL TRIAL: NCT06676878
Title: Assessment of Differences in Body Composition, Physical Fitness, and Thermoregulatory Response to Incremental Exercise in Young Boys With Type I Diabetes and Healthy Soccer Players
Brief Title: Body Composition, Fitness, and Thermoregulation in Young Boys With Type I Diabetes vs. Healthy Soccer Players
Acronym: BCFTYR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Paweł Korman (Other)
Responsible Party: Sponsor-Investigator, Paweł Korman, Assistant professor, Poznan University of Physical Education
Organization: Poznan University of Physical Education (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 654/24
Record Dates: First submitted 2024-10-20; First posted 2024-11-06 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Diabetes
Keywords: diabetes; football; exercise; thermography
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes (Experimental): The study group will consist exclusively of diabetics and they will undergo the described treadmill stress test to exhaustion.
  Interventions: Device: Incremental exercise
- Control (Active Comparator): The control group will consist exclusively of healthy participants and they will undergo the described treadmill stress test to exhaustion (identical to the study group).
  Interventions: Device: Incremental exercise

INTERVENTIONS:
Device: Incremental exercise — A graded exercise test will be performed on a treadmill. After 3 minutes of standing on the treadmill, participants will walk at a speed of 4 km/h for the first 3 minutes, then the speed will be increased to 8 km/h. After this point, the treadmill speed will be increased by 2 km/h every 3 minutes until voluntary exhaustion.

SUMMARY:
The study aims to assess differences in body composition, exercise capacity, and thermoregulation between young soccer players with type 1 diabetes and their healthy peers. Real-time glycemic monitoring during exercise will provide insights for developing effective diabetes management strategies, enhancing athletes' health and performance.

DETAILED DESCRIPTION:
The aim of the study is to assess differences in body composition, exercise capacity, and exercise-induced thermoregulation between young athletes (soccer players) with type 1 diabetes and their healthy peers (also soccer players). Specifically, the study seeks to understand how type 1 diabetes, periodic glycemic fluctuations, and the body's metabolic balance status impact these parameters. By monitoring glycemic levels in real-time during exercise, the research will provide valuable insights into the necessity and frequency of glycemic control for individuals engaging in physical activity of varying intensities. The data obtained from this study may be crucial for developing effective strategies for managing type 1 diabetes in athletes, ultimately contributing to the improvement of their overall health and physical performance. Additionally, these findings could inform guidelines and recommendations for safe and effective exercise practices for diabetic athletes.

ELIGIBILITY:
Inclusion Criteria:

* Active soccer training for at least 5 years

Exclusion Criteria:

* Comorbidities significantly affecting metabolism and thermoregulation

Ages: 15 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-08-26 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Skin temperature changes | during the test
  Thermal images of the lower limbs will be taken using a thermal camera (Flir SC 640, manufactured in the USA) before, during, and after exercise (during recovery). The assessment will be performed in degrees Celsius (°C).
Core temperature changes | Core temperature recording will start 12 hours before the exercise test and continue throughout its duration.
  Core temperature will be measured using the eCelsius Performance system (BodyCap, France).

SECONDARY OUTCOMES:
Glycemic monitoring | during the test
  Athletes with type 1 diabetes (study group) and healthy individuals (control group) will also have a continuous glucose monitoring sensor (FreeStyle Libra, Abbott Medical, Warsaw, Poland, or similar) placed on the back of one arm. The sensors will be applied one week before the exercise test and will remain active for 14 days. Glucose levels will be measured in milligrams per deciliter (mg/dL).

OTHER OUTCOMES:
Antropometric measurement - weight | before test
  Body weight (kg) will be measured using a digital stadiometer (SECA 285, SECA, Hamburg, Germany).
Antropometric measurement - height | before test
  Body height (cm) will be measured using a digital stadiometer (SECA 285, SECA, Hamburg, Germany).
Bone Mineral Density (BMD): | before test
  Bone Mineral Density (BMD) will be measured using dual-energy X-ray absorptiometry (DXA) with the Lunar Prodigy Pro DXA device (GE Healthcare, Madison, WI, USA) and enCORE v. 16 SP1 software. BMD is expressed in grams per square centimeter (g/cm²) and indicates the density of minerals, such as calcium, in bones. All DXA scans will be performed and analyzed by the same trained technician according to the manufacturer's protocols to ensure consistency and accuracy. The procedure involves the participant lying on a table while a low-dose X-ray scans their body. The process is non-invasive and generally considered safe, with minimal exposure to radiation, comparable to the amount received during a cross-country flight.
Fat Mass | before test
  Fat Mass will be assessed using the DXA method with the Lunar Prodigy Pro DXA device and enCORE v. 16 SP1 software. This parameter is measured in kilograms (kg) or as a percentage of total body weight (%), representing the total mass of fat in the body.All DXA scans will be performed and analyzed by the same trained technician according to the manufacturer's protocols to ensure consistency and accuracy. The procedure involves the participant lying on a table while a low-dose X-ray scans their body. The process is non-invasive and generally considered safe, with minimal exposure to radiation, comparable to the amount received during a cross-country flight.
Lean Mass | before test
  Lean Mass will also be measured using the DXA method. This includes the weight of muscles, organs, and other non-fat tissues, expressed in kilograms (kg). All DXA scans will be performed and analyzed by the same trained technician according to the manufacturer's protocols to ensure consistency and accuracy. The procedure involves the participant lying on a table while a low-dose X-ray scans their body. The process is non-invasive and generally considered safe, with minimal exposure to radiation, comparable to the amount received during a cross-country flight.
Ventilation | during test
  Ventilation will be measured using an ergospirometer (Cortex Metamax 3B R2, Leipzig, Germany) and analyzed with MetasoftStudio v. 5.1.0 software (Cortex-Metamax 3B R2; Cortex Biophysik, Leipzig, Germany). The ventilation parameter will be expressed in liters per minute (L/min), which allows for the assessment of the volume of air inhaled and exhaled by the participant per minute.
Oxygen Consumption (VO2) | during the test
  Oxygen consumption (VO2) will be measured using an ergospirometer (Cortex Metamax 3B R2, Leipzig, Germany) and analyzed with MetasoftStudio v. 5.1.0 software (Cortex-Metamax 3B R2; Cortex Biophysik, Leipzig, Germany). The VO2 parameter will be expressed in milliliters per kilogram per minute (mL/kg/min), which allows for the assessment of the amount of oxygen consumed by the body per unit of body weight per minute.
Measurement Cardiovascular Parameters | during the test
  A Polar Bluetooth Smart HR H6 heart rate monitor (Polar Electro Oy, Kempele, Finland) will be used to monitor heart rate (HR), measured in beats per minute (bpm).
Monitoring Fatigue Levels Using the RPE Scale | during the test
  The Rating of Perceived Exertion (RPE) scale will be used to monitor fatigue levels during exercise. The RPE will be measured on a scale from 6 to 20.
  Level 6 on the RPE scale indicates no exertion. This is the lowest level, suggesting that the exercise requires no physical effort.
  Level 20 on the RPE scale indicates maximum exertion. This is the highest level, suggesting that the exercise is performed with the maximum possible effort, at the limit of endurance.
Lactate | during the test
  To measure lactate accumulation, a Biosen C-line (EKF Diagnostics, Barleben, Germany) will be used. In brief, 20 µL of whole blood will be drawn into a prefilled micro test tube using a capillary. The L-lactate contained in the sample will be enzymatically converted to pyruvate and hydrogen peroxide, which will be detected by the electrode. The lactate concentration will be measured in mmol/L.
Glucose Levels from a Fingertip Blood Drop | during the test
  To measure glucose levels, a glucose meter (e.g., Accu-Chek, Roche Diagnostics, Mannheim, Germany) will be used. In brief, a small drop of blood will be obtained from the fingertip using a lancet. The blood sample will then be placed on a test strip inserted into the glucose meter. The glucose in the sample will react with the chemicals on the strip, producing an electrical signal that will be measured by the meter. The glucose concentration will be displayed in mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Straburzynska-Lupa, Prof, Study Director — Department of Physical Therapy and Sports Recover, Poznan University of Physical Education
Locations (1):
- Human Movement Analysis Laboratory LaBthletics Academy of Physical Education in Poznań, Poznan, Wlkp, Poland

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be disclosed except for information that allows for the personal identification of study participants.
Supporting Information: Study Protocol, ICF
Time Frame: 09.2025 - 12.2026
Access Criteria: Access to Individual Participant Data (IPD) is granted to researchers affiliated with recognized academic or healthcare institutions for legitimate scientific research purposes.

REFERENCES:
- [Background] Wierzbicka E, Swiercz A, Pludowski P, Jaworski M, Szalecki M. Skeletal Status, Body Composition, and Glycaemic Control in Adolescents with Type 1 Diabetes Mellitus. J Diabetes Res. 2018 Sep 3;2018:8121634. doi: 10.1155/2018/8121634. eCollection 2018. PMID 30250851
- [Background] Mysliwiec A, Skalska M, Michalak A, Chrzanowski J, Szmigiero-Kawko M, Lejk A, Jastrzebska J, Radziminski L, Lopez-Sanchez GF, Gawrecki A, Jastrzebski Z. Responses to Low- and High-Intensity Exercise in Adolescents with Type 1 Diabetes in Relation to Their Level of VO2 Max. Int J Environ Res Public Health. 2021 Jan 15;18(2):692. doi: 10.3390/ijerph18020692. PMID 33467392
- [Background] De Ridder F, Ledeganck KJ, De Winter B, Braspenning R, Delbeke D, Renard E, Pozzilli P, Pieralice S, Vissers D, De Block C. Trends of glucose, lactate and ketones during anaerobic and aerobic exercise in subjects with type 1 diabetes: The ACTION-1 study. Diabetes Metab Res Rev. 2022 Sep;38(6):e3537. doi: 10.1002/dmrr.3537. Epub 2022 May 21. PMID 35533265
- [Background] Reddy R, Wittenberg A, Castle JR, El Youssef J, Winters-Stone K, Gillingham M, Jacobs PG. Effect of Aerobic and Resistance Exercise on Glycemic Control in Adults With Type 1 Diabetes. Can J Diabetes. 2019 Aug;43(6):406-414.e1. doi: 10.1016/j.jcjd.2018.08.193. Epub 2018 Aug 30. PMID 30414785
- [Background] McGinn R, Carter MR, Barrera-Ramirez J, Sigal RJ, Flouris AD, Kenny GP. Does type 1 diabetes alter post-exercise thermoregulatory and cardiovascular function in young adults? Scand J Med Sci Sports. 2015 Oct;25(5):e504-14. doi: 10.1111/sms.12344. Epub 2014 Dec 8. PMID 25487370
- Available data/document: Study Protocol — https://drive.google.com/file/d/1q_WKKHXRUchhM8gDnu0EHNJ1AU-UH4M4/view?usp=drive_link
- Available data/document: Informed Consent Form — https://drive.google.com/file/d/1q_WKKHXRUchhM8gDnu0EHNJ1AU-UH4M4/view?usp=drive_link

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2026-01-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT06676878/Prot_ICF_001.pdf